CLINICAL TRIAL: NCT06867744
Title: Extracapsular Supradiscal Subperiosteal Surgical Procedure for Temporomandibular Joint Internal Derangement Correction: Novel Technique''
Brief Title: Extracapsular Supradiscal Subperiosteal Surgical Procedure for Temporomandibular Joint Internal Derangement Correction: Novel Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Moawed Ibrahim Ghoneim, PhD (Other)
Collaborators: Menoufia University (Other); Sinai University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Moawed Ibrahim Ghoneim, PhD, Associate professor, Sinai University
Organization: Sinai University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS 1-10-023
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: TMJ Internal Derangement; TMJ - Dislocation of Temporomandibular Joint; TMJ - Oral &Maxillofacial Surgery
Keywords: TMJ; TMJ derangement; extracapsular surgery; supradiscal subperiosteal technique; facial plastic surgery

STUDY DESIGN:
Intervention Model Description: A prospective study was conducted on 50 patients (47 females, 3 males; age range: 11-50 years) with TMJ ID refractory to non-surgical management. The ESS procedure was performed to reposition the displaced disc and stabilize retrodiscal tissues without violating the joint capsule. Preoperative and postoperative assessments included pain levels, maximum mouth opening (MMO), and subjective patient feedback
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temporomandibular Joint Internal Derangement Correction (Other): The ESS procedure was performed to reposition the displaced disc and stabilize retrodiscal tissues without violating the joint capsule. Preoperative and postoperative assessments included pain levels, maximum mouth opening (MMO), and subjective patient feedback.
  Interventions: Procedure: Extracapsular Supradiscal Subperiosteal Surgical Procedure for Temporomandibular Joint Internal Derangement Correction

INTERVENTIONS:
Procedure: Extracapsular Supradiscal Subperiosteal Surgical Procedure for Temporomandibular Joint Internal Derangement Correction — Patients in a supine extended position with nasotracheal intubation; oral intubation in such cases is not suitable as it makes dissection and disc repositioning difficult and compromises the surgery results. Periauricular incision with postauricular extension; after infiltration with noradrenaline 1/200000 solution with or without zylocaine which gives better exposure and better aesthetic results. Dissection down the wound till reach the temporal fascia starting posteriorlay till the fascia blended with the zygomatic arch anteriorly; identification of temporal root of zygomatic arch using fine dissector followed by subperiosteal dissection of zygomatic arch till five mm anterior to the articular eminence of TMJ. Accurate identification of TMJ followed by meticulous subperiosteal dissection of superior margin of TMJ capsule then the dissection continued posteriorly till posterior margin; no need to dissect the bilaminar zone, and the dissection continued anteriorly down the skull base t

SUMMARY:
This study aims to evaluate the efficacy of the ESS technique in correcting TMJ internal derangement, with a focus on functional outcomes and patient satisfaction.

DETAILED DESCRIPTION:
Background: Internal derangement (ID) of the temporomandibular joint (TMJ) is a prevalent condition characterized by disc displacement, leading to pain, restricted mandibular mobility, and reduced quality of life. While non-surgical treatments are often the first line of management, surgical intervention becomes necessary in refractory cases. Traditional surgical methods, such as arthrocentesis and disc repositioning, have shown variable success rates, particularly in advanced stages of disc damage. This study introduces the Extracapsular Supradiscal Subperiosteal (ESS) surgical procedure, a novel technique designed to address these limitations. Therefore, current study aims to evaluate the efficacy of the ESS technique in correcting TMJ internal derangement, with a focus on functional outcomes and patient satisfaction.

Patients and Methods: A prospective study was conducted on 50 patients (47 females, 3 males; age range: 11-50 years) with TMJ ID refractory to non-surgical management. The ESS procedure was performed to reposition the displaced disc and stabilize retrodiscal tissues without violating the joint capsule. Preoperative and postoperative assessments included pain levels, maximum mouth opening (MMO), and subjective patient feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 3 or stage 4 internal derangements of TMJ radiological and clinical findings should coincide to set up the diagnosis and predict the treatment plan.

Exclusion Criteria:

* Age less than 11 years old
* Age more than 50 years are excluded

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
TMJ Pain | 3 months
  change of pain on a visual analogue scale (VAS) from 0 to 10 with decreased number means less pain
Interincisal Distance Score | pre- and post operative (3 days)
  Interincisal Distance Scores from score-0 to score-3 to be identified
Jaw deviation during Mouth Opening | 3 days
  A 13-score evaluating the jaw deviation during mouth opening from score-0 to score-12
Clicking | 3 months
  The clicking during mouth opening scores among study participants, both pre- and postoperative
HIT-6 | 3 days
  the Headache impact test (HIT-6) both pre- and postoperatively among study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Faculty of Medicine, University Hospital, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
A prospective study was conducted on 50 patients (47 females, 3 males; age range: 11-50 years) with TMJ ID refractory to non-surgical management. The ESS procedure was performed to reposition the displaced disc and stabilize retrodiscal tissues without violating the joint capsule. Preoperative and postoperative assessments included pain levels, maximum mouth opening (MMO), and subjective patient feedback.